CLINICAL TRIAL: NCT03147677
Title: A Prospective, Multi-center, Randomized, Open-label, Parallel-arm Controlled Study of Treating Type 2 Diabetic Nephropathy (Stage II-IV) With Alfacalcidol and Irbesartan
Brief Title: Clinical Study of Treating Type 2 Diabetic Nephropathy With Alfacalcidol and Irbesartan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 320.6750.16025
Record Dates: First submitted 2017-04-06; First posted 2017-05-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetic Nephropathy
Keywords: Type 2 diabetic nephropathy; Alfacalcidol
MeSH Terms: interventions — alfacalcidol; Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alfacalcidol and Irbesartan (Experimental): The subjects in this group orally take Alfacalcidol Soft Capsules at 0.25ug/day and Irbesartan Pills at 150mg/day for 16 consecutive weeks.All subjects will be followed up for 4 weeks after medication is over. A total of 4 visits have been scheduled for this study at week 0, week 8, week 16, week 20.
  Interventions: Drug: Alfacalcidol; Drug: Irbesartan
- Irbesartan (Active Comparator): The subjects in this group orally take Irbesartan Pills at 150mg/day for 16 consecutive weeks.All subjects will be followed up for 4 weeks after medication is over. A total of 4 visits have been scheduled for this study at week 0, week 8, week 16, week 20.
  Interventions: Drug: Irbesartan
- Alfacalcidol (Active Comparator): The subjects in this group orally takeAlfacalcidol Soft Capsules at 0.25ug/day for 16 consecutive weeks.All subjects will be followed up for 4 weeks after medication is over. A total of 4 visits have been scheduled for this study at week 0, week 8, week 16, week 20.
  Interventions: Drug: Alfacalcidol

INTERVENTIONS:
Drug: Alfacalcidol
  Other Names: Alfacalcidol Soft Capsules
  Arms: Alfacalcidol; Alfacalcidol and Irbesartan
Drug: Irbesartan
  Other Names: Irbesartan Pills
  Arms: Alfacalcidol and Irbesartan; Irbesartan

SUMMARY:
This is a prospective, multi-center, randomized, open-label, parallel-arm controlled study, for which a total of 216 patients with type 2 diabetic nephropathy (Stage II-IV) will be enrolled. The subjects will be randomized to three groups in 1:1:1 ratio. One group receive Alfacalcidol 0.25ug/day and Irbesartan 150mg/day for 16 consecutive weeks. The second group receive Alfacalcidol 0.25ug/day alone for 16 consecutive weeks. The third group receive Irbesartan 150mg/day alone for 16 consecutive weeks. All subjects will be followed up for 4 weeks after medication is over. A total of 4 visits have been scheduled for this study at week 0, week 8, week 16, week 20.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chinese subjects, at age 18-65, diagnosed with Type 2 diabetic nephropathy (Stage II-IV) who meet the WHO diagnostic standards of diabetes in 1999. The international Mogensen staging standard for diabetic nephropathy is used. Specifically, in Stage II (normal albuminuria stage), the UAER is normal (<20μg /min or<30mg/24h). In Stage III (early diabetic nephropathy stage), the UAER is 20-200μg /min or 30-300 mg/24h. In Stage IV (clinical or overt diabetic nephropathy stage), the UAER is >200μg/min or urine protein quantitation is >500mg /24h.

Exclusion Criteria:

* Renal damage caused by other causes;
* Uncontrolled hypertension (blood pressure constantly greater than 140/ 90mmHg);
* Type 1 Diabetes
* Any acute and chronic infections;
* Glycosylated hemoglobin (HbA1c)>7.5%;
* 24h urinary protein quantity>3g, serum albumin<25g /L and estimated glomerular filtration rate (eGFR)<60 ml/min;
* Patients who suffered from malignant tumors or any illness that endanger life, such as liver, kidney, heart and lung function insufficiency over the past 5 years;
* People who have received the gastrointestinal operation, which may affect absorption of Vitamin D;
* People who have taken such drugs as angiotensin receptor blocker, calcium, and angiotensin converting enzyme inhibitor that affect excretion of urine protein, and who have been allergic to Vitamin D;
* Pregnant or lactating women;
* Other candidates that are deemed not suitable by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in 24h urinary albumin excretion rate (UAER) by comparing visits at week 20 with the baseline | at Week 20
Changes in 24h urinary protein quantity by comparing visits at week 20 with the baseline | at Week 20

SECONDARY OUTCOMES:
Changes in estimated glomerular filtration rate (eGFR) by comparing visits at week 20 with the baseline | at Week 20
Changes in the urine levels of IL-6, MCP-1, TGF-β1, MIP-1β, and PTPN2 by comparing visits at week 20 with the baseline. | at Week 20
Changes in serum levels of IL-6, MCP-1, TGF-β1, MIP-1β, and PTPN2 by comparing visits at week 20 with the baseline. | at Week 20
Changes in urinary albumin / creatinine (UACR) of morning urine by comparing visits at week 20 with the baseline | at Week 20

OTHER OUTCOMES:
Incidence of all adverse events (AEs) and serious adverse events (SAEs) | during the whole study from week 0 to week 20

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zhang, Doctor, Study Chair — The Third Xiangya Hospital of Central South University
Locations (3):
- China (3):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Chenzhou NO.1 People's Hospital, Chenzhou, Hunan
  - Hunan Yiyang Central Hospital, Yiyang, Hunan

IPD SHARING:
Plan to Share IPD: No